CLINICAL TRIAL: NCT05439304
Title: RoboCare - Implementation of a Smart Robot in Care Homes
Brief Title: RoboCare - Technology in Care Homes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: The Dam Foundation (Other); Norwegian Health Association (Other)
Responsible Party: Sponsor
Other Study IDs: 401080
Record Dates: First submitted 2022-06-14; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Dementia
Keywords: Care home; Technology; Person centred care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Care staff
  Interventions: Other: No intervention
- Residents
  Interventions: Other: No intervention
- Family members
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study primary objective of this study is to identify promoting and hindering factors that affect the implementation of a smart robot in a care home setting.

DETAILED DESCRIPTION:
People living with dementia represents a vulnerable group with a high need for person centred care to maintain a high quality of life. Loneliness and social isolation is already a common problem in care homes and has become a global challenge during the pandemic because of its negative effect on health. As a response to missing social interactions, technology with the intent to enhance communication and encourage activities have been introduced in care homes. However, there is a lack of knowledge about the introduction and use of technology. To gain insight into this, Centre for Age-Related Medicine at Stavanger University Hospital SESAM has carried out a pilot project made possible by DAM Foundation, where the smart robot Berntsen (hereinafter referred to as Berntsen) was used for video communication. The pilot project show that the use requires organizational leadership, motivated care staff and a well-organized introduction, and that there is a great need for more knowledge about these factors in order to develop a good implementation strategy.

Hence, SESAM has started the ground breaking project "RoboCare - Effectiveness, efficiency, uptake and use of a smart robot in care homes: A cluster randomized trial and implementation study" to investigate if Berntsen can reduce loneliness and social isolation, increase residents' quality of life and increase staff job satisfaction. Berntsen is an iPad on a stand with wheels or a tripod suitable for tabled tops, with content that can be customized to the user. It can promote person centred activities, tailored schedules and facilitate video communication. Berntsen can also act as a personal trainer with customized exercise videos in collaboration with a physical therapist.

This study will be part of the cluster RCT to explore which factors are important for implementation from the micro-level (person with dementia, family member and staff) perspective, and what must be set for optimal use of Berntsen in a care home.

It is of vital importance that all stakeholders are involved in an implementation process to integrate technology. These aspects are however less described in research concerning development of technological interventions in care homes. Consequently, knowledge concerning care staff, residents and informal carers is scarce.

Design: An explorative qualitative study consisting of 3 sub studies:

1. A qualitative study to investigate the resident, family member and care staff perspective on implementation and use of technology in a care home setting
2. A qualitative study to investigate the resident, family member and care staff experience using Berntsen as part of daily practice and for communication.
3. A qualitative observational study to investigate the dynamic between people living with dementia and family member during communication through Berntsen.

ELIGIBILITY:
Care staff:

* Any care staff in the included care homes will be invited to participate

Residents

Inclusion Criteria:

* Dementia diagnosis at the time of inclusion equivalent with stage 5 (Moderately severe cognitive decline) on the Functional Assessment Staging Tool (FAST)

Exclusion Criteria:

* Any participants who are not able to give informed consent themselves or through a consultee will not be included in the project.

Family member

* All family members of included residents will be invited to participate in the project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from two care homes also included in the cluster RCT. For diversity purposes, we seek to include both large and smaller care homes from larger cities and rural areas and purposely include two different units from each care to reflect the variety of experiences.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hindering and promoting factors to technology implementation | Three years
  Measured using qualitative interviews with care staff, residents and family members and observation of residents and family members

SECONDARY OUTCOMES:
Implementation and use of technology in a care home setting | July - December 2022
  Measured by qualitative focus group interviews with care staff, and individual interviews with residents and family members in dyads. Interviews will be based on semi-structured interview guide.
User perspective on Berntsen | January - June 2023
  Measured by qualitative focus group interviews with care staff, and individual interviews with residents and family members in dyads. Interviews will be based on semi-structured interview guide.
People with dementia and family member communication through Berntsen | July - December 2023
  Measured by observation of people living with dementia and family members during communication through Berntsen. Observations will be based on an observation guide.

REFERENCES:
- [Background] Ballard C, Corbett A, Orrell M, Williams G, Moniz-Cook E, Romeo R, Woods B, Garrod L, Testad I, Woodward-Carlton B, Wenborn J, Knapp M, Fossey J. Impact of person-centred care training and person-centred activities on quality of life, agitation, and antipsychotic use in people with dementia living in nursing homes: A cluster-randomised controlled trial. PLoS Med. 2018 Feb 6;15(2):e1002500. doi: 10.1371/journal.pmed.1002500. eCollection 2018 Feb. PMID 29408901
- [Background] Barbosa Neves B, Sanders A, Kokanovic R. "It's the worst bloody feeling in the world": Experiences of loneliness and social isolation among older people living in care homes. J Aging Stud. 2019 Jun;49:74-84. doi: 10.1016/j.jaging.2019.100785. Epub 2019 Jun 6. PMID 31229221
- [Background] Ko M, Wagner L, Spetz J. Nursing Home Implementation of Health Information Technology: Review of the Literature Finds Inadequate Investment in Preparation, Infrastructure, and Training. Inquiry. 2018 Jan-Dec;55:46958018778902. doi: 10.1177/0046958018778902. PMID 29888677
- [Background] Khosravi P, Ghapanchi AH. Investigating the effectiveness of technologies applied to assist seniors: A systematic literature review. Int J Med Inform. 2016 Jan;85(1):17-26. doi: 10.1016/j.ijmedinf.2015.05.014. Epub 2015 Jun 11. PMID 26216463